CLINICAL TRIAL: NCT04683523
Title: Anaerobic Exercise Impact on Cardiac Workload, Peripheral Resistance and Lipid Index Among Grade 1 HTN Patients
Brief Title: Anaerobic Exercises on Cardiac Workload, Peripheral Resistance and Lipid Index Among Grade 1 Hypertensive Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Ali Farhad, Assistant professor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ziauddin U
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaerobic exercise training (Experimental)
  Interventions: Other: Exercise
- Aerobic exercise training (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Resistance training using dumbbells and therabands

SUMMARY:
Impact of resistance exercises on grade I hypertensive patients were monitored on three outcome measures that were blood pressure, peripheral resistance and lipid index after 12 weeks of intervention

ELIGIBILITY:
Inclusion Criteria:

* grade I HTN Age 20-40years Both male and female

Exclusion Criteria:

* unable to perform exercises Comorbidities like Diabetes

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | From baseline to 12 weeks of training
  Sphygmomanometer
Peripheral Resistance | From baseline to 12 weeks of training
  Ankle Brachial Index
Lipid index | From baseline to 12 weeks of intervention
  Hdl to ldl ratio blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Farhad, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No